CLINICAL TRIAL: NCT06101251
Title: A Randomized Field Trial of Smartphone-based Feedback Designed to Encourage Safe Driving: Comparing Focused and Self-chosen Goals to Standard UBI Messaging
Brief Title: A Randomized Field Trial of Smartphone-based Feedback to Encourage Safe Driving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: AAA Foundation for Traffic Safety (Unknown)
Responsible Party: Principal Investigator, M. Kit Delgado, MD, Assistant Professor of Emergency Medicine and Epidemiology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 853761
Record Dates: First submitted 2023-07-27; First posted 2023-10-26 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Distracted Driving; Injury Prevention; Behavioral Economics
Keywords: Distracted Driving; Behavioral Incentives

STUDY DESIGN:
Intervention Model Description: At the end of the 6-week baseline period, participants who have the app installed and collecting data, and who meet a minimum number of driver trips with trips scores, will be randomized into one of 4 arms via Way to Health:
  Arm 1, Control: Way to Drive app only monitors trips in the background
  Arm 2, Standard feedback + UBI-like Financial Incentive: Receive weekly feedback on all four behaviors and overall driver safety; safety tips on all four behaviors; up to $100 based on their overall driver safety at end of intervention.
  Arm 3, Assigned Goal + UBI-like Financial Incentive: Receive weekly feedback on behavior that presents greatest opportunity for improvement; safety tips on this behavior; up to $100 based on their overall driver safety at end of intervention.
  Arm 4, Self-Chosen Goal + UBI-like Financial Incentive: Receive weekly feedback on behavior of their own choosing; safety tips on this behavior; up to $100 based on their overall driver safety at end of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Participants will have the Way to Drive app monitoring in the background throughout the intervention period for overall driving score, handheld phone use, speeding, hard braking, and fast acceleration. They will not receive feedback, driving tips or UBI-like behavioral incentives.
  Participants will also receive payment or non-adherence messages as needed for having the app functioning.
- Standard Feedback + UBI-like Behavioral Incentive (Active Comparator): Participants will have the Way to Drive app monitoring in the background, and will receive payment or non-adherence messages as needed, but will also receive, Standard Feedback, Study Dashboard, Driving Tips, and UBI-like Behavioral Incentive
  Interventions: Behavioral: Driving Tips; Behavioral: Standard Feedback; Behavioral: Study Dashboard (Standard); Behavioral: UBI-like Behavioral Incentive
- Assigned Goal with UBI-like Behavioral Incentive (Active Comparator): Participants will have the Way to Drive app monitoring in the background, and will receive payment or non-adherence messages as needed, but will also receive Assigned Focus Area Feedback, Driving Tips, a Study Dashboard, and UBI-like Behavioral Incentive
  Interventions: Behavioral: Driving Tips; Behavioral: Assigned Focus Area Feedback; Behavioral: Study Dashboard (focused); Behavioral: UBI-like Behavioral Incentive
- Self-Chosen Goal with UBI-like Behavioral Incentive (Active Comparator): Participants will have the Way to Drive app monitoring in the background, and will receive payment or non-adherence messages as needed, but will also receive Self-Chosen Focus Area Feedback, Driving Tips, Study Dashboard, and UBI-like Behavioral Incentive.
  Interventions: Behavioral: Driving Tips; Behavioral: Study Dashboard (Standard); Behavioral: UBI-like Behavioral Incentive; Behavioral: Sef-Chosen Focus Area Feedback

INTERVENTIONS:
Behavioral: Driving Tips — Each week participants will receive a safe driving tip for one of the four behaviors via text message.
  Arms: Assigned Goal with UBI-like Behavioral Incentive; Self-Chosen Goal with UBI-like Behavioral Incentive; Standard Feedback + UBI-like Behavioral Incentive
Behavioral: Standard Feedback — Each week participants will receive a text message showing their overall driving score (out of 100) and subscores for distraction, hard braking, fast acceleration, and speeding (all running averages). The scoreboard will indicate whether their scores have gone up, down, or stayed the same. The message will include a link to a dashboard.
  Arms: Standard Feedback + UBI-like Behavioral Incentive
Behavioral: Assigned Focus Area Feedback — Each week feedback will focus the participant's attention on the driving behavior with the greatest opportunity for improvement based on their baseline driving behavior. Participants will be assigned a goal for the week of a score 5 points (3 points in the case of Driver Focus) better than their baseline for that area. If they meet the goal, they will be given a new goal 5 points higher; if they fall short, they will be asked to try for the same goal again. If they improve sufficiently-or if their improvement stalls out-they will be assigned a new behavior to focus on.
  Arms: Assigned Goal with UBI-like Behavioral Incentive
Behavioral: Study Dashboard (Standard) — By clicking the link in the feedback text, they will be able to view a weekly dashboard that provides detailed information about their baseline, best, last, and average scores for each of the four behaviors, plus descriptions of the four behaviors.
  Arms: Self-Chosen Goal with UBI-like Behavioral Incentive; Standard Feedback + UBI-like Behavioral Incentive
Behavioral: Study Dashboard (focused) — Same as standard study dashboard, except participants will see at the top of the dashboard how well they are doing relative to their weekly goals.
  Arms: Assigned Goal with UBI-like Behavioral Incentive
Behavioral: UBI-like Behavioral Incentive — At the end of the 12-week intervention period, their overall driving score will be translated into a $0-$100 reward amount. For example, a participant with an overall driving score of 84 at the end of the intervention period would receive $84 in compensation.
  Arms: Assigned Goal with UBI-like Behavioral Incentive; Self-Chosen Goal with UBI-like Behavioral Incentive; Standard Feedback + UBI-like Behavioral Incentive
Behavioral: Sef-Chosen Focus Area Feedback — Participants will be asked to select which driving behavior they want to focus on improving, and to set a goal for the week that is above their baseline score. If they meet the goal, they will be asked to set a new, higher goal; if they fall short, they will be asked to try for the same goal again. If they improve sufficiently-or if their improvement stalls out-they will be asked if they want to focus on a new behavior.
  Arms: Self-Chosen Goal with UBI-like Behavioral Incentive

SUMMARY:
The study team are proposing to conduct a randomized controlled trial to determine the effectiveness of focused feedback vs standard feedback and self-chosen vs assigned goals on driving behaviors targeted by behavior-based insurance apps: hard braking, fast acceleration, handheld phone use, and speeding. The interventions arms will receive feedback on their driving behaviors, tips for safe driving, and a UBI-like financial incentive. The Penn research team will use Meta advertisements to recruit for the study and determine eligibility via an online survey. Those who enroll will undergo a 6-week run-in period during which their driving trips will be monitored by a mobile app. Individuals with a sufficient number of trips during this period will be randomly assigned to one of four arms for the intervention period. Target enrollment is 1,300 participants (325 per trial arm). The power analysis assumed an attrition rate of 20% over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Has an Apple or Android smartphone (iPhone iOS 12 or later or Android OS 7 or later)
* Drives at least 2 days per week
* English reading ability
* Passes an attention check
* Provides valid email address, cell number, name, address, and date of birth

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1449 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Overall Driving Score | 12 weeks of the intervention period + separate analysis of 6 week post intervention.
  This is the mean of the four behavior scores for the intervention period (and, in a follow-up analysis of effect sustainability, the post-intervention period). Scores can range from 0 -100, 100 being the safest driving score.

SECONDARY OUTCOMES:
Distraction score | 12 weeks of the intervention period + separate analysis of 6 week post intervention.
  A proprietary CMT score based on participant phone use-especially handheld phone use-while driving on a scale of 0-100, 100 being no phone use while driving (safest).
Speeding score | 12 weeks of the intervention period + separate analysis of 6 week post intervention.
  A proprietary CMT score based on the amount of time the participant drove over the speed limit on a scale from 0 -100, 100 being no incidences of driving over the speed limit.
Braking score | 12 weeks of the intervention period + separate analysis of 6 week post intervention.
  A proprietary CMT score based on the frequency of a participant's hard brakes on a scale of 0-100, 100 meaning no hard brakes.
Acceleration Score | 12 weeks of the intervention period + separate analysis of 6 week post intervention.
  A proprietary CMT score based on the frequency of a participant's fast accelerations on a scale of 0-100. 100, being no fast accelerations.

OTHER OUTCOMES:
Handheld phone use per hour of driving | 12 weeks of the intervention period + separate analysis of 6 week post intervention.
  This is a composite outcome that measures the proportion of total trip time in which the driver is engaged in handheld phone call use or non-call handheld use (e.g. texting, swiping, and typing), as measured by the Way to Drive app. Several studies (e.g. Klauer, NEJM, 2014) have demonstrated the association between handheld phone use (e.g., reaching for phone, typing, swiping, dialing) and increased crash risk. This outcome is also known as the active phone use percentage. Passive phone use (e.g. phone is streaming GPS navigation directions or music without any typing, swiping, or holding of the phone) is not included in this outcome.
Overall riskiness metric | 12 weeks of the intervention period + separate analysis of 6 week post intervention.
  This is a composite measure of the underlying driving metrics for the four behaviors of interest. For each behavior a z-score will be computed for each participant and take the mean of these four z-scores to get their overall riskiness. This will be done for both the intervention period and the post-intervention period.
Disabled SMS messaging | 18 weeks of the study (6 - week baseline; 12- week intervention period)
  If a participant texts "stop" or "bye" to stop receiving our intervention text messages, this could indicate unacceptability of push notification interventions. This will be measured as a binary score, where participants that text "stop" or "bye" will be marked as 1, and those that do not will be marked as 0.
Unenrolled | 18 weeks of the study (6 - week baseline; 12- week intervention period)
  If a participant asks to be unenrolled, this is an even stronger indicator of unacceptability. This will be measured as a binary score, where 1 means the participant was unenrolled before the end of the intervention period, and 0 means they were not.
Net Promoter Score (NPS) | At 24 weeks.
  This will be derived for each arm based on a 1-item question on a scale of 0 -10, 0 bring not at all likely to recommend the program, and 10 being extremely likely.
4-item acceptability scale | At 24 weeks.
  This will be a 4-item acceptability scale administered in the exit survey. For each participant the mean of the 4 items will be calculated for an overall acceptability score ranging from 1-5 (5 is the best).
Intervention helpfulness. | At 24 weeks.
  Intervention arm participants will be asked to rate the helpfulness of each of the 4 intervention components (SMS feedback, weekly dashboard, SMS tips, $100 incentive), each on a scale of 1 (not at all) to 5 (extremely), with an option to indicate they did not see or were not aware of the intervention component.
Hard braking events per 100 miles of driving | 12 weeks of the intervention period + separate analysis of 6 week post intervention.
  Number of hard braking evens per 100 miles of driving
Minutes of speeding per hour of driving. | 12 weeks of the intervention period + separate analysis of 6 week post intervention.
  Based on duration of speeding events detected by the app.
Fast acceleration events per 100 miles of driving. | 12 weeks of the intervention period + separate analysis of 6 week post intervention.
  Number of fast acceleration events per 100 miles of driving.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States